CLINICAL TRIAL: NCT03020212
Title: Long-term Oxygen Therapy in Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Live at High Altitude (2640 Meters Above Sea Level): Evaluation of a Proposal for Adjusting Criteria
Brief Title: Long-term Oxygen Therapy in Patients With Chronic Obstructive Pulmonary Disease Who Live at High Altitude
Acronym: COPD-LTOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Neumologica Colombiana (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COLP
Record Dates: First submitted 2016-05-13; First posted 2017-01-13 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease; High altitude; Oxygen; long-term oxygen therapy; pulmonary hypertension; chronic hypoxemia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Altitude Sickness; Hypertension, Pulmonary | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Active Comparator): Long-term oxygen therapy in patients with chronic obstructive pulmonary disease (COPD)
  Interventions: Drug: Oxygen
- Not oxygen (No Intervention): No intervention ( no therapy with oxygen)

INTERVENTIONS:
Drug: Oxygen — The subjects will be randomly assigned to receive or not LTOT and they will be followed for 30 months. At baseline and then at 10, 20 and 30 months, they will be clinically evaluated with arterial blood gases, pulse oximetry, echocardiography, spirometry with bronchodilator, diffusion capacity, quality of life (SGRQ), neurocognitive performance (MMSE) and six minutes walk test. The primary outcome will evaluate the ratio of occurrence of erythrocytosis or pulmonary hypertension. Secondary outcomes will be evaluated quality of life, lung function, neurocognitive performance and exercise tolerance by comparing the groups with and without LTOT.
  Other Names: LTOT
  Arms: Oxygen

SUMMARY:
A clinical, prospective, randomized controlled trial to determine the effect of prescribing oxygen in a group of COPD (chronic pulmonary disease) patients with PaO2 (arterial oxygen tension) ≥50 and ≤55 mmHg who do not have erythrocytosis or pulmonary hypertension on echocardiogram (which are considered manifestations of chronic hypoxia)

DETAILED DESCRIPTION:
A clinical, prospective, randomized controlled trial to determine the effect of prescribing oxygen in a group of COPD patients with PaO2 ≥50 and ≤55 mmHg who do not have erythrocytosis or pulmonary hypertension on echocardiogram (which are considered manifestations of chronic hypoxia). It will be included 220 patients of the Fundación Neumológica Colombiana living in Bogotá who accept their participation by signing an informed consent.

The subjects will be randomly assigned to receive or not LTOT and they will be followed for 20 to 30 months. At baseline and then at 10, 20 and 30 months, they will be clinically evaluated with arterial blood gases, pulse oximetry, echocardiography, spirometry with bronchodilator, diffusion capacity, quality of life (SGRQ), neurocognitive performance (MMSE) and six minutes walk test. The primary outcome will evaluate the ratio of occurrence of erythrocytosis or pulmonary hypertension. Secondary outcomes will be evaluated quality of life, lung function, neurocognitive performance and exercise tolerance by comparing the groups with and without LTOT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ≥ 40 years and < 85 years living in Bogotá or in a high - altitude city (>2.500 - <3.500 m).
* Diagnosis of COPD defined by FEV1 / FVC <LLN (Lower limit of normal value) and significant exposure to cigarette ≥ 10 packs / year or woodsmoke ≥ 10 years.
* Diagnosis of ACO defined by FEV1 / FVC post BD <70%, significant exposure to cigarette or woodsmoke and asthma diagnosed before 40 years and/or wheezing, cough with spirometry with a high respond to bronchodilator (FEV1 or FVC ≥ 15% and 400 ml) or eosinophil >300 cels.
* PaO2 ≥ 50 and ≤ 55 mmHg or oxygen desaturation during the six-minute walk test (at least in three of the measurements performed during the exam) or during sleep (SpO2 ≤ 85% in ≥ 30% of the total time of sleep)
* No clinical signs of cor pulmonale
* Clinically stable COPD defined as no exacerbations in the last three months.
* Signature of informed consent.

Exclusion Criteria:

* BMI ≥40.
* Paraclinical findings of chronic hypoxemia and pulmonary hypertension:

  * Hematocrit ≥ 55%.
  * Pulmonary hypertension (PH) defined by transthoracic echocardiography systolic pulmonary artery pressure > 40 mmHg or indirect signs of PH: Pulmonary artery acceleration time <100ms associated with a meso-systolic notch and flattening of the septum interventricular in systole.
* Echocardiographic findings that could lead to pulmonary hypertension.

  * Left ventricular systolic dysfunction defined by an ejection fraction <40%
  * Left ventricular diastolic dysfunction higher than grade I.
  * Valvular disease higher than moderate
* Use of oxygen > 12 hours a day for more than six months in the last year.
* Comorbidities not controlled or deemed medically that can contribute to mortality during the study follow-up.
* Diagnosis of severe sleep apnea-hypopnea syndrome without treatment
* Plan of transfer of residence below 2.500 meters.
* Medical, psychiatric, social and administrative conditions that define high probability of poor adherence to therapy with oxygen.
* Active smoking

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-02; Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Development of pulmonary hypertension | 3 years
  An echocardiogram will be conducted every ten months to measure the value of pulmonary artery pressure and establish the presence of pulmonary hypertension

SECONDARY OUTCOMES:
Development of polycythemia | 3 years
  A sample of hematocrit and hemoglobine will be perfomed to establish the presence of polycythemia at the begining of the study and every 10 months.
Evaluation of the pulmonary function | 3 years
  Spirometry will be conducted to assess the Forced expiratory volume at 1 second and the Forced vital capacity at the begining of the study and every 10 months.
Number of exacerbations | 3 years
  It will report the number of exacerbations that present the patients during the study
Evaluation of the quality of life | 3 years
  It will perform the St. George Respiratory Questionnaire (SGRQ) to assess the quality of life of the patients at the begining of the study and every 10 months.
Assessment of neurocognitive function | 3 years
  It will make a Mini mental Test to evaluate the neurocognitive performance at the begining of the study and every 10 months.
Evaluation of exercise tolerance | 3 years
  It will conduct a six minute walk test to assess the exercise tolerance at the the begining of the study and every 10 months.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Torres-Duque, MD, Principal Investigator — Fundación Neumológica Colombiana
Locations (1):
- Fundación Neumológica Colombiana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim V, Benditt JO, Wise RA, Sharafkhaneh A. Oxygen therapy in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2008 May 1;5(4):513-8. doi: 10.1513/pats.200708-124ET. PMID 18453364
- [Background] Montes de Oca M, Lopez Varela MV, Acuna A, Schiavi E, Rey MA, Jardim J, Casas A, Tokumoto A, Torres Duque CA, Ramirez-Venegas A, Garcia G, Stirbulov R, Camelier A, Bergna M, Cohen M, Guzman S, Sanchez E. ALAT-2014 Chronic Obstructive Pulmonary Disease (COPD) Clinical Practice Guidelines: questions and answers. Arch Bronconeumol. 2015 Aug;51(8):403-16. doi: 10.1016/j.arbres.2014.11.017. Epub 2015 Jan 14. English, Spanish. PMID 25596991
- [Background] Diaz-Lobato S, Mayoralas Alises S. [Should we reconsider the criteria for home oxygen therapy depending on altitude?]. Arch Bronconeumol. 2011 Aug;47(8):421-2. doi: 10.1016/j.arbres.2011.05.001. Epub 2011 Jul 6. No abstract available. Spanish. PMID 21737196
- [Background] Semenza GL. HIF-1: mediator of physiological and pathophysiological responses to hypoxia. J Appl Physiol (1985). 2000 Apr;88(4):1474-80. doi: 10.1152/jappl.2000.88.4.1474. PMID 10749844
- [Background] Mannino DM, Buist AS. Global burden of COPD: risk factors, prevalence, and future trends. Lancet. 2007 Sep 1;370(9589):765-73. doi: 10.1016/S0140-6736(07)61380-4. PMID 17765526
- [Background] Pauwels RA, Rabe KF. Burden and clinical features of chronic obstructive pulmonary disease (COPD). Lancet. 2004 Aug 14-20;364(9434):613-20. doi: 10.1016/S0140-6736(04)16855-4. PMID 15313363
- [Background] Hurd S. The impact of COPD on lung health worldwide: epidemiology and incidence. Chest. 2000 Feb;117(2 Suppl):1S-4S. doi: 10.1378/chest.117.2_suppl.1s. PMID 10673465
- [Background] Murray CJ, Lopez AD. Global mortality, disability, and the contribution of risk factors: Global Burden of Disease Study. Lancet. 1997 May 17;349(9063):1436-42. doi: 10.1016/S0140-6736(96)07495-8. PMID 9164317
- [Background] Safe S, Hutzinger O, Ecobichon DJ, Grey AA. The metabolism of 4'chloro-4-biphenylol in the rat. Can J Biochem. 1975 Apr;53(4):415-20. doi: 10.1139/o75-057. PMID 1125825
- [Background] Barbera JA, Peinado VI, Santos S. Pulmonary hypertension in chronic obstructive pulmonary disease. Eur Respir J. 2003 May;21(5):892-905. doi: 10.1183/09031936.03.00115402. PMID 12765440
- [Background] Hu J, Discher DJ, Bishopric NH, Webster KA. Hypoxia regulates expression of the endothelin-1 gene through a proximal hypoxia-inducible factor-1 binding site on the antisense strand. Biochem Biophys Res Commun. 1998 Apr 28;245(3):894-9. doi: 10.1006/bbrc.1998.8543. PMID 9588211
- [Background] Hochachka PW. Mechanism and evolution of hypoxia-tolerance in humans. J Exp Biol. 1998 Apr;201(Pt 8):1243-54. doi: 10.1242/jeb.201.8.1243. PMID 9510535
- [Background] Juel C, Lundby C, Sander M, Calbet JA, Hall Gv. Human skeletal muscle and erythrocyte proteins involved in acid-base homeostasis: adaptations to chronic hypoxia. J Physiol. 2003 Apr 15;548(Pt 2):639-48. doi: 10.1113/jphysiol.2002.035899. Epub 2003 Feb 28. PMID 12611920
- [Background] McClelland GB, Brooks GA. Changes in MCT 1, MCT 4, and LDH expression are tissue specific in rats after long-term hypobaric hypoxia. J Appl Physiol (1985). 2002 Apr;92(4):1573-84. doi: 10.1152/japplphysiol.01069.2001. PMID 11896024
- [Background] McDonald CF, Blyth CM, Lazarus MD, Marschner I, Barter CE. Exertional oxygen of limited benefit in patients with chronic obstructive pulmonary disease and mild hypoxemia. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 1):1616-9. doi: 10.1164/ajrccm.152.5.7582304.
- [Background] Weitzenblum E, Chaouat A, Kessler R. Long-term oxygen therapy: do current guidelines need revision? Eur Respir J. 1999 May;13(5):1209-10. doi: 10.1034/j.1399-3003.1999.13e44.x. No abstract available. PMID 10414428
- [Background] Hardinge M, Annandale J, Bourne S, Cooper B, Evans A, Freeman D, Green A, Hippolyte S, Knowles V, MacNee W, McDonnell L, Pye K, Suntharalingam J, Vora V, Wilkinson T; British Thoracic Society Home Oxygen Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guidelines for home oxygen use in adults. Thorax. 2015 Jun;70 Suppl 1:i1-43. doi: 10.1136/thoraxjnl-2015-206865. PMID 25870317
- [Result] Katsenos S, Constantopoulos SH. Long-Term Oxygen Therapy in COPD: Factors Affecting and Ways of Improving Patient Compliance. Pulm Med. 2011;2011:325362. doi: 10.1155/2011/325362. Epub 2011 Sep 15. PMID 21941649
- [Result] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Result] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Result] Caballero A, Torres-Duque CA, Jaramillo C, Bolivar F, Sanabria F, Osorio P, Orduz C, Guevara DP, Maldonado D. Prevalence of COPD in five Colombian cities situated at low, medium, and high altitude (PREPOCOL study). Chest. 2008 Feb;133(2):343-9. doi: 10.1378/chest.07-1361. Epub 2007 Oct 20. PMID 17951621
- [Result] Menezes AM, Perez-Padilla R, Jardim JR, Muino A, Lopez MV, Valdivia G, Montes de Oca M, Talamo C, Hallal PC, Victora CG; PLATINO Team. Chronic obstructive pulmonary disease in five Latin American cities (the PLATINO study): a prevalence study. Lancet. 2005 Nov 26;366(9500):1875-81. doi: 10.1016/S0140-6736(05)67632-5. PMID 16310554
- [Result] Yu AY, Frid MG, Shimoda LA, Wiener CM, Stenmark K, Semenza GL. Temporal, spatial, and oxygen-regulated expression of hypoxia-inducible factor-1 in the lung. Am J Physiol. 1998 Oct;275(4):L818-26. doi: 10.1152/ajplung.1998.275.4.L818. PMID 9755115
- [Result] Casanova C, Celli BR, Barria P, Casas A, Cote C, de Torres JP, Jardim J, Lopez MV, Marin JM, Montes de Oca M, Pinto-Plata V, Aguirre-Jaime A; Six Minute Walk Distance Project (ALAT). The 6-min walk distance in healthy subjects: reference standards from seven countries. Eur Respir J. 2011 Jan;37(1):150-6. doi: 10.1183/09031936.00194909. Epub 2010 Jun 4. PMID 20525717
- [Result] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Result] Garina IA, Rakitskaya VV, Shalyapina VG. Receptor binding of corticosterone in monoaminergic structures of the brain of rats after neonatal blockade of the hypophyseoadrenal system. Neurosci Behav Physiol. 1991 Sep-Oct;21(5):387-90. doi: 10.1007/BF01200271. No abstract available. PMID 1758616
- [Result] Casanova C, Cote C, Marin JM, Pinto-Plata V, de Torres JP, Aguirre-Jaime A, Vassaux C, Celli BR. Distance and oxygen desaturation during the 6-min walk test as predictors of long-term mortality in patients with COPD. Chest. 2008 Oct;134(4):746-752. doi: 10.1378/chest.08-0520. Epub 2008 Jul 14. PMID 18625667
- [Result] Hiraga T, Maekura R, Okuda Y, Okamoto T, Hirotani A, Kitada S, Yoshimura K, Yokota S, Ito M, Ogura T. Prognostic predictors for survival in patients with COPD using cardiopulmonary exercise testing. Clin Physiol Funct Imaging. 2003 Nov;23(6):324-31. doi: 10.1046/j.1475-0961.2003.00514.x. PMID 14617262
- [Result] Drummond MB, Blackford AL, Benditt JO, Make BJ, Sciurba FC, McCormack MC, Martinez FJ, Fessler HE, Fishman AP, Wise RA; NETT Investigators. Continuous oxygen use in nonhypoxemic emphysema patients identifies a high-risk subset of patients: retrospective analysis of the National Emphysema Treatment Trial. Chest. 2008 Sep;134(3):497-506. doi: 10.1378/chest.08-0117. Epub 2008 Jul 18. PMID 18641094
- [Result] Stein DA, Bradley BL, Miller WC. Mechanisms of oxygen effects on exercise in patients with chronic obstructive pulmonary disease. Chest. 1982 Jan;81(1):6-10. doi: 10.1378/chest.81.1.6. No abstract available. PMID 6797795
- [Result] Hardinge M, Suntharalingam J, Wilkinson T; British Thoracic Society. Guideline update: The British Thoracic Society Guidelines on home oxygen use in adults. Thorax. 2015 Jun;70(6):589-91. doi: 10.1136/thoraxjnl-2015-206918. Epub 2015 Apr 27. PMID 25918120